CLINICAL TRIAL: NCT00147602
Title: A Double-Blind, Randomized, Placebo- Controlled Study Of Atorvastatin As Prevention Of Cerebrovascular Events In Patients With A Previous Transient Ischemic Attack (TIA) Or Stroke
Brief Title: Lipitor In The Prevention Of Stroke, For Patients Who Have Had A Previous Stroke
Acronym: SPARCL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0981-342; A2581138
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Atorvastatin

INTERVENTIONS:
Drug: atorvastatin

SUMMARY:
To determine whether Lipitor reduces stroke, compared to placebo in patients who have had a previous stroke or transient ischemic attack.

ELIGIBILITY:
Inclusion Criteria:

* Previous stroke or TIA

Exclusion Criteria:

* coronary heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4732
Dates: Start 1998-11; Study Completion 2005-11

PRIMARY OUTCOMES:
Time to occurrence of fatal or non-fatal stroke

SECONDARY OUTCOMES:
Time to occurrence of an acute coronary event, consisting of cardiac death, nonfatal myocardial infarction, resuscitated cardiac arrest or unstable angina.
Time to occurrence of a cerebrovascular event, defined as fatal or nonfatal stroke or TIA.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (118):
- Australia (7):
  - Pfizer Investigational Site, East Gosford, New South Wales
  - Pfizer Investigational Site, Randwick, Sydney, New South Wales
  - Pfizer Investigational Site, Footscray, Victoria
  - Pfizer Investigational Site, Heidelberg Heights, Victoria
  - Pfizer Investigational Site, Parkville, Victoria
  - Pfizer Investigational Site, Prahran, Victoria
  - Pfizer Investigational Site, Perth, Western Australia
- Austria (4):
  - Pfizer Investigational Site, Graz
  - Pfizer Investigational Site, Innsbruck
  - Pfizer Investigational Site, Vienna
  - Pfizer Investigational Site, Villach
- Belgium (4):
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Tielt
  - Pfizer Investigational Site, Waregem
- Brazil (2):
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Pfizer Investigational Site, Viña del Mar, Chile
- Czechia (6):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Ostrava
  - Pfizer Investigational Site, Ostrava-Poruba
  - Pfizer Investigational Site, Pilsen
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Zlín
- Denmark (3):
  - Pfizer Investigational Site, Copenhagen Nv
  - Pfizer Investigational Site, Glostrup Municipality
  - Pfizer Investigational Site, Hellerup
- Finland (6):
  - Pfizer Investigational Site, Hus, Helsinki
  - Pfizer Investigational Site, Kotka
  - Pfizer Investigational Site, Kuopio
  - Pfizer Investigational Site, Lahti
  - Pfizer Investigational Site, Lappeenranta
  - Pfizer Investigational Site, Oulu
- France (8):
  - Pfizer Investigational Site, Saint-Denis, Cedex 1
  - Pfizer Investigational Site, Paris, Cedex 20
  - Pfizer Investigational Site, Toulouse, Cedex 3
  - Pfizer Investigational Site, Bourg-en-Bresse, Cedex
  - Pfizer Investigational Site, Besançon
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Paris
- Germany (10):
  - Pfizer Investigational Site, Bad Rodach
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Mannheim
  - Pfizer Investigational Site, Minden
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Münster
  - Pfizer Investigational Site, Regensburg
- Greece (3):
  - Pfizer Investigational Site, Athens, Melissia
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Thessaloniki
- Israel (4):
  - Pfizer Investigational Site, Haifa
  - Pfizer Investigational Site, Holon
  - Pfizer Investigational Site, Petah Tikva
  - Pfizer Investigational Site, Tel Aviv
- Italy (6):
  - Pfizer Investigational Site, Via Brunamonti 15, Perugia
  - Pfizer Investigational Site, Bari
  - Pfizer Investigational Site, Bergamo
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Monza
- Pfizer Investigational Site, Monterrey, Nuevo León, Mexico
- Netherlands (6):
  - Pfizer Investigational Site, Rotterdam, Gelderland
  - Pfizer Investigational Site, Almelo
  - Pfizer Investigational Site, Delft
  - Pfizer Investigational Site, Goes
  - Pfizer Investigational Site, RB Groningen
  - Pfizer Investigational Site, Tilburg
- New Zealand (3):
  - Pfizer Investigational Site, Takapuna, Auckland
  - Pfizer Investigational Site, Auckland
  - Pfizer Investigational Site, Christchurch
- Poland (7):
  - Pfizer Investigational Site, Bialystok
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Sosnowiec
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- Portugal (3):
  - Pfizer Investigational Site, Coimbra Codex
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Porto
- Pfizer Investigational Site, Bratislava, Slovakia
- South Africa (3):
  - Pfizer Investigational Site, Bloemfontein
  - Pfizer Investigational Site, Cape Town
  - Pfizer Investigational Site, Parow
- Spain (11):
  - Pfizer Investigational Site, Alicante, Alicante
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, L'Hospitalet (bcn), Barcelona
  - Pfizer Investigational Site, Burgos, Burgos
  - Pfizer Investigational Site, Girona, Girona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, MÃ¡laga, Malaga
  - Pfizer Investigational Site, Seville, Sevilla
  - Pfizer Investigational Site, Valencia, Valencia
  - Pfizer Investigational Site, Zaragoza, Zaragoza
  - Pfizer Investigational Site, Palma de Mallorca
- Sweden (5):
  - Pfizer Investigational Site, Danderyd
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Umeå
  - Pfizer Investigational Site, Uppsala
  - Pfizer Investigational Site, Västervik
- Switzerland (5):
  - Pfizer Investigational Site, Aarau
  - Pfizer Investigational Site, Basel
  - Pfizer Investigational Site, Bern
  - Pfizer Investigational Site, Lausanne
  - Pfizer Investigational Site, Zurich
- United Kingdom (8):
  - Pfizer Investigational Site, Dundee, Scotland
  - Pfizer Investigational Site, Newport, South Wales
  - Pfizer Investigational Site, Aberdeen
  - Pfizer Investigational Site, Cardiff
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Liverpool
  - Pfizer Investigational Site, Nottingham
  - Pfizer Investigational Site, Woolwich
- Pfizer Investigational Site, Caracas, Venezuela

REFERENCES:
- [Result] Amarenco P, Bogousslavsky J, Callahan A 3rd, Goldstein LB, Hennerici M, Rudolph AE, Sillesen H, Simunovic L, Szarek M, Welch KM, Zivin JA; Stroke Prevention by Aggressive Reduction in Cholesterol Levels (SPARCL) Investigators. High-dose atorvastatin after stroke or transient ischemic attack. N Engl J Med. 2006 Aug 10;355(6):549-59. doi: 10.1056/NEJMoa061894. PMID 16899775
- [Derived] Chemello K, Gallo A, Guedon AF, Techer R, Croyal M, Swietek MJ, Meilhac O, Amarenco P, Lambert G. Lipoprotein(a): A Residual Cardiovascular Risk Factor in Statin-Treated Stroke Survivors: Insights From the SPARCL Trial. JACC Adv. 2023 Aug 22;2(7):100557. doi: 10.1016/j.jacadv.2023.100557. eCollection 2023 Sep. PMID 38939496
- [Derived] Szarek M, Amarenco P, Callahan A, DeMicco D, Fayyad R, Goldstein LB, Laskey R, Sillesen H, Welch KM; SPARCL Committees and Investigators. Atorvastatin Reduces First and Subsequent Vascular Events Across Vascular Territories: The SPARCL Trial. J Am Coll Cardiol. 2020 May 5;75(17):2110-2118. doi: 10.1016/j.jacc.2020.03.015. Epub 2020 Mar 16. PMID 32194196
- [Derived] Vogt L, Bangalore S, Fayyad R, Melamed S, Hovingh GK, DeMicco DA, Waters DD. Atorvastatin Has a Dose-Dependent Beneficial Effect on Kidney Function and Associated Cardiovascular Outcomes: Post Hoc Analysis of 6 Double-Blind Randomized Controlled Trials. J Am Heart Assoc. 2019 May 7;8(9):e010827. doi: 10.1161/JAHA.118.010827. PMID 31020900
- [Derived] Ganz P, Amarenco P, Goldstein LB, Sillesen H, Bao W, Preston GM, Welch KMA; SPARCL Steering Committee. Association of Osteopontin, Neopterin, and Myeloperoxidase With Stroke Risk in Patients With Prior Stroke or Transient Ischemic Attacks: Results of an Analysis of 13 Biomarkers From the Stroke Prevention by Aggressive Reduction in Cholesterol Levels Trial. Stroke. 2017 Dec;48(12):3223-3231. doi: 10.1161/STROKEAHA.117.017965. Epub 2017 Nov 7. PMID 29114094
- [Derived] Byun YS, Yang X, Bao W, DeMicco D, Laskey R, Witztum JL, Tsimikas S; SPARCL Trial Investigators. Oxidized Phospholipids on Apolipoprotein B-100 and Recurrent Ischemic Events Following Stroke or Transient Ischemic Attack. J Am Coll Cardiol. 2017 Jan 17;69(2):147-158. doi: 10.1016/j.jacc.2016.10.057. PMID 28081824
- [Derived] Amarenco P, Callahan A 3rd, Campese VM, Goldstein LB, Hennerici MG, Messig M, Sillesen H, Welch KM, Wilson DJ, Zivin JA. Effect of high-dose atorvastatin on renal function in subjects with stroke or transient ischemic attack in the SPARCL trial. Stroke. 2014 Oct;45(10):2974-82. doi: 10.1161/STROKEAHA.114.005832. Epub 2014 Aug 21. PMID 25147328
- [Derived] Ovbiagele B, Goldstein LB, Amarenco P, Messig M, Sillesen H, Callahan A 3rd, Hennerici MG, Zivin J, Welch KM; SPARCL Investigators. Prediction of major vascular events after stroke: the stroke prevention by aggressive reduction in cholesterol levels trial. J Stroke Cerebrovasc Dis. 2014 Apr;23(4):778-84. doi: 10.1016/j.jstrokecerebrovasdis.2013.12.001. Epub 2014 Feb 24. PMID 24582273
- [Derived] Callahan A, Amarenco P, Goldstein LB, Sillesen H, Messig M, Samsa GP, Altafullah I, Ledbetter LY, MacLeod MJ, Scott R, Hennerici M, Zivin JA, Welch KM; SPARCL Investigators. Risk of stroke and cardiovascular events after ischemic stroke or transient ischemic attack in patients with type 2 diabetes or metabolic syndrome: secondary analysis of the Stroke Prevention by Aggressive Reduction in Cholesterol Levels (SPARCL) trial. Arch Neurol. 2011 Oct;68(10):1245-51. doi: 10.1001/archneurol.2011.146. Epub 2011 Jun 13. PMID 21670382
- [Derived] Schwartz GG, Chaitman BR, Goldberger JJ, Messig M. High-dose atorvastatin and risk of atrial fibrillation in patients with prior stroke or transient ischemic attack: analysis of the Stroke Prevention by Aggressive Reduction in Cholesterol Levels (SPARCL) trial. Am Heart J. 2011 May;161(5):993-9. doi: 10.1016/j.ahj.2011.02.002. PMID 21570534
- [Derived] Amarenco P, Goldstein LB, Sillesen H, Benavente O, Zweifler RM, Callahan A 3rd, Hennerici MG, Zivin JA, Welch KM; Stroke Prevention by Aggressive Reduction in Cholesterol Levels Investigators. Coronary heart disease risk in patients with stroke or transient ischemic attack and no known coronary heart disease: findings from the Stroke Prevention by Aggressive Reduction in Cholesterol Levels (SPARCL) trial. Stroke. 2010 Mar;41(3):426-30. doi: 10.1161/STROKEAHA.109.564781. Epub 2010 Jan 28. PMID 20110538
- [Derived] Amarenco P, Goldstein LB, Callahan A 3rd, Sillesen H, Hennerici MG, O'Neill BJ, Rudolph AE, Simunovic L, Zivin JA, Welch KM; SPARCL Investigators. Baseline blood pressure, low- and high-density lipoproteins, and triglycerides and the risk of vascular events in the Stroke Prevention by Aggressive Reduction in Cholesterol Levels (SPARCL) trial. Atherosclerosis. 2009 Jun;204(2):515-20. doi: 10.1016/j.atherosclerosis.2008.09.008. Epub 2008 Sep 18. PMID 18962621